CLINICAL TRIAL: NCT05857995
Title: Precision Lung Cancer Survivorship Care Intervention: A Randomized Controlled Trial Serving Rural Survivors and Communities
Brief Title: Precision Lung Cancer Survivorship Care Intervention
Acronym: KYLEADSII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jerod L Stapleton, PhD (Other)
Collaborators: University of Louisville (Other); G02 for Lung Cancer (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jerod L Stapleton, PhD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 94571; R01CA254734 (NIH)
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer; Pulmonary Neoplasm; Neoplasms, Lung; Neoplasms, Pulmonary; Neoplasm, Pulmonary; Cancer, Lung; Cancers, Lung; Pulmonary Cancer; Cancer, Pulmonary; Cancers, Pulmonary; Pulmonary Cancers; Cancer of the Lung; Cancer of Lung; Pulmonary Neoplasms; Lung Cancers
Keywords: Survivorship; Quality of Life; Behavioral Oncology; Psychosocial Oncology
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Two-group randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigators and outcomes assessors will be masked to the random assignment of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kentucky LEADS Collaborative Lung Cancer Survivorship Care Program (KLCLCSC) (Experimental): The Kentucky LEADS Collaborative Lung Cancer Survivorship Care Program (KLCLCSC) is a targeted and tailored lung cancer survivorship care intervention built on principles of patient-centered care, shared decision making, and motivational interviewing to build survivor engagement and improve lung cancer outcomes.
  Interventions: Behavioral: Kentucky LEADS Collaborative Lung Cancer Survivorship Care Program
- Enhanced Usual Care (EUC) (Active Comparator): The enhanced usual care condition involves usual care plus bibliotherapy and assessment.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Kentucky LEADS Collaborative Lung Cancer Survivorship Care Program — KLCLCSC is a survivor or survivor plus caregiver-focused psychosocial and behavioral intervention designed to engage lung cancer survivors and improve lung cancer outcomes.
  Arms: Kentucky LEADS Collaborative Lung Cancer Survivorship Care Program (KLCLCSC)
Behavioral: Enhanced Usual Care — EUC involves a combination of the standard of care plus a bibliotherapy intervention and assessment.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The overarching goal of the Kentucky LEADS Collaborative Lung Cancer Survivorship Care program is to reduce the burden of lung cancer by offering an innovative survivorship care approach that improves lung cancer quality of life, overcomes lung cancer stigma, and helps survivors engage with care. The project involves a two-group parallel randomized clinical trial comparing the impact of the Kentucky LEADS Collaborative Lung Cancer Survivorship Care program (KLCLCSC) among lung cancer survivors (N=300) against an enhanced usual care condition (bibliotherapy+assessment) on quality of life outcomes.

DETAILED DESCRIPTION:
Among the devastating illnesses impacting rural America, few exact the physical, social, psychological, and economic toll of lung cancer. Lung cancer is the leading cause of cancer death in rural America, and the levy is particularly acute in Kentucky - a state that not only leads the nation in lung cancer incidence and mortality but is a global epicenter of lung cancer. Despite the prevailing nihilism regarding lung cancer care, lung cancer survivors are living longer. Innovations in prevention, early detection, and treatment, have created substantial optimism and opportunities for long-term lung cancer survivorship. These dramatic changes in the lung cancer care landscape have invigorated the need for quality lung cancer survivorship interventions. The overarching goal of the Kentucky LEADS Collaborative Lung Cancer Survivorship Care program is to reduce the burden of lung cancer by offering an innovative survivorship care approach that improves lung cancer quality of life, overcomes lung cancer stigma, and helps survivors engage with care. Using a novel precision survivorship approach and developed in collaboration with rural community stakeholders, the program's foundation incorporates principles of patient-centered care, shared decision making, and motivational interviewing to build survivor engagement. A large acceptability and feasibility trial conducted in collaboration with nine lung cancer care facilities in Kentucky with lung cancer survivors (N=140) demonstrated the acceptability of the intervention among survivors, caregivers, and lung cancer care clinicians. The study also revealed the feasibility of conducting the proposed study methods in rural cancer care facilities. The project continues this program of research by conducting a two-group parallel randomized clinical trial comparing the impact of the Kentucky LEADS Collaborative Lung Cancer Survivorship Care program (KLCLCSC) among lung cancer survivors (N=300) against an enhanced usual care condition (bibliotherapy+assessment) on quality of life outcomes. Rural-residing lung cancer survivors will be recruited from ten oncology care facilities throughout Kentucky. The project's first aim compares the efficacy of the interventions with regard to lung cancer quality of life among survivors as measured by the FACT-L and other rigorous assessments of patient engagement, symptom burden, psychosocial well-being, and behavior change. The project's second aim evaluates the moderating impact of including caregivers as intervention partners on survivor quality of life outcomes. A third aim evaluates the cost-effectiveness of the KLCLCSC intervention in comparison to the enhanced usual care condition. Based on highly encouraging pilot data collected in collaboration with oncology care programs in Kentucky, this research holds credible potential to establish a new paradigm for addressing the challenges associated with lung cancer and for delivering quality survivorship care to rural-residing, economically distressed lung cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with lung cancer
* Reside in a rural county as determined by a Rural Urban Continuum Code (RUC) of 4 or higher
* Be at least 18 years of age or older
* Be able to communicate effectively in English

Exclusion Criteria:

* Have significant psychiatric disturbance that requires a higher level of care
* Have substance abuse/dependence that requires a higher level of care
* Are participating in another lung cancer survivorship care intervention
* Have previously participated in the Kentucky LEADS Lung Cancer Survivorship Care Program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline (T0) in Mean Lung Cancer Quality of Life at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  The Functional Assessment of Cancer Therapy-Lung (FACT-L) is a 36-item self-report instrument that measures quality life. Scores range from 0 to 144 with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Change from Baseline (T0) in Total Survivor Engagement at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  The Patient Activation Measure (PAM) is a standardized 13-item self-report measure of patient engagement with a theoretical range of 0 to 100 with higher scores indicating greater engagement.
Change from Baseline (T0) in Mean Lung Cancer Knowledge at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  The Perceived Knowledge of Lung Cancer Scale is a 6-item intervention-specific measure of self-reported/perceived knowledge of lung cancer and survivorship developed for this research program. Scores range from 0 to 24 with higher scores indicating greater knowledge.
Change from Baseline (T0) in Mean Fatigue Symptoms at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  Fatigue Symptoms is a standardized 5-item self-report measure of fatigue within the Patient-Reported Outcomes Measurement Information System (PROMIS-Fatigue). Scores range from 0 to 20 with higher scores indicating better quality of life and lesser fatigue symptoms.
Change from Baseline (T0) in Mean Sleep Disturbance at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  Sleep Disturbance is a standardized 6-item self-report measure of sleep disruption within the Patient-Reported Outcomes Measurement Information System (PROMIS-Sleep). Scores range from 0 to 20 with higher scores indicating better quality of life and lesser seep disturbance.
Change from Baseline (T0) in Pulmonary Symptoms at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  Respiratory Dysfunction (FACT-L Pulmonary Symptom Index) is a 4-item self-report measure of breathing problems drawn from the Functional Assessment of Cancer Therapy Lung Cancer Module. Scores range from 0 to 16 with higher scores indicating better quality of life and lower pulmonary symptoms.
Change from Baseline (T0) in Mean Pain Interference at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  Pain Interference is a standardized 6-item self-report measure of pain interference within the Patient-Reported Outcomes Measurement Information System (PROMIS-Pain). Scores range from 0 to 24 with higher scores indicating better quality of life and lesser pain interference.
Change from Baseline (T0) in Mean Emotional Social Support at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  Emotional Social Support is a standardized 4-item self-report measure of emotional social support within the Patient-Reported Outcomes Measurement Information System (PROMIS-Emotional Support). Scores range from 0 to 16 with higher scores indicating better quality of life and greater emotional social support.
Change from Baseline (T0) in Mean Knowledge of Palliative Care at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  The Knowledge of Palliative Care (Perceptions) scale is a standardized 4-item self-report measure of knowledge about palliative care. Scores range from 4 to 16 with higher scores indicating greater self-rated knowledge of palliative care.
Change from Baseline (T0) in Psychological Distress at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  The Distress Thermometer is an ultra-brief, single-item, standardized self-report measure of psychological distress developed and supported by the National Comprehensive Cancer Network (DT) with higher scores indicating greater distress (Range = 0 to 10).
Change from Baseline (T0) in Mean Physical Activity at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  The Godin Leisure-Time Exercise Questionnaire includes 3 standardized self-report items assessing levels of strenuous, moderate, and mild/light physical activity. Scores are based on weekly activities with zero being the lowest score and higher scores indicating more frequent and strenuous physical activity.
Change from Baseline (T0) in Smoking Status at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  The Smoking Status (BRFSS-Tobacco Use) measure is a single-item standardized self-report measure of 30-day smoking point prevalence. Scores range from 0 to 1 with 1 indicating current smoking.
Change from Baseline (T0) in Lung Cancer Stigma at 6 Months (T2) | Baseline (T0) and 6 Months (T2)
  The Lung Cancer Stigma Inventory - Short Form includes 12 self-report items measuring lung cancer stigma. Scores range from 12 to 60 with higher scores indicating greater lung cancer stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Studts, PhD, Principal Investigator — University of Colorado School of Medicine; Jerod L Stapleton, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No